CLINICAL TRIAL: NCT04329312
Title: Differential Diagnosis of Pulmonary Hypertension With Automated Image Analysis - a Pilot Study
Brief Title: Differential Diagnosis of Pulmonary Hypertension With Automated Image Analysis
Status: Terminated | Type: Observational
Why Stopped: slow recruitment
Sponsor: Medical University of Graz (Other)
Collaborators: Ludwig Boltzmann Institute for Lung Vascular Research (Other)
Responsible Party: Sponsor
Other Study IDs: 32-184 ex 19/20
Record Dates: First submitted 2020-03-30; First posted 2020-04-01 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- Pulmonary arterial hypertension (PAH): The patients with PAH received an invasive right-heart catheterization and a thoracic CT scan as part of their routine work up.
  Interventions: Radiation: Thoracic computed tomography
- PH due to left-heart disease (PH-LHD): The patients with PH-LHD received an invasive right-heart catheterization and a thoracic CT scan as part of their routine work up.
  Interventions: Radiation: Thoracic computed tomography
- Chronic thromboembolic pulmonary hypertension (CTEPH): The patients with CTEPH received an invasive right-heart catheterization and a thoracic CT scan as part of their routine work up.
  Interventions: Radiation: Thoracic computed tomography
- PH due to emphysema (PH-LD-Emphys): The patients with PH-LD-Emphys received an invasive right-heart catheterization and a thoracic CT scan as part of their routine work up.
  Interventions: Radiation: Thoracic computed tomography
- PH due to lung fibrosis (PH-LD-Fibr): The patients with PH-LD-Fibr received an invasive right-heart catheterization and a thoracic CT scan as part of their routine work up.
  Interventions: Radiation: Thoracic computed tomography
- PH due to combined emphysema and fibrosis (PH-LD-CPFE): The patients with PH-LD-CPFE received an invasive right-heart catheterization and a thoracic CT scan as part of their routine work up.
  Interventions: Radiation: Thoracic computed tomography
- No PH: The patients without PH received an invasive right-heart catheterization and a thoracic CT scan as part of their routine work up.
  Interventions: Radiation: Thoracic computed tomography

INTERVENTIONS:
Radiation: Thoracic computed tomography — Patients undergo contrast-enhanced thoracic computed tomography as part of their routine clinical work up.

SUMMARY:
The aim of the study is to determine relevant morphologic parameters of the lung vasculature for the differentiation between different groups of patients with pulmonary hypertension (PH) by thoracic computer tomography (CT). In this pilot study patients undergoing right heart catheterization will be investigated by thoracic CT and special software to determine morphologic readouts.

The investigators expect that using this non-invasive method, parameters relevant for the differentiation of the patients with PH can be determined.

DETAILED DESCRIPTION:
Pulmonary hypertension (PH) is defined as an elevated mean pressure in the pulmonary artery above 20mmHg determined at right-heart catheterization. Depending on the presentation and pathogenesis, patients are classified according to five main groups. A correct classification is crucial, since it is essential for the available therapy options.

A promising non-invasive method to provide important hemodynamic and clinical Information is the fully-automatic analysis of thoracic computed tomography images. This method can yield a number of quantitative morphologic readouts of the lung vasculature and the parenchyma.

This study aims to identify quantitative markers from the fully-automatic image analysis, which allow a discrimination between the various PH patient groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients with right-heart catheterization
* Clinical indication for thoracic CT

Exclusion Criteria:

* Pregnancy
* Decreased kidney function
* Intolerance to contrast material
* Other standard CT contraindications

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Populations are recruited from the patients visiting the outpatient clinic for pulmonology of the Medical University of Graz.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Lung vessel morphology | 1 day
  Quantitative measures of lung vessel morphology based on automated CT image analysis based on artery-vein separation and vessel segmentation, which allow differentiation between the different groups of PH

CONTACTS AND LOCATIONS:
Overall Officials: Horst Olschewski, MD, Principal Investigator — Medical University of Graz
Locations (1):
- Medical University Graz, Division of Pulmonology, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: No